CLINICAL TRIAL: NCT00566566
Title: Adipocytokines as Predictors of the Metabolic Syndrome in Survivors of Childhood Acute Lymphoblastic Leukemia
Brief Title: Adipokines as Predictors of the Metabolic Syndrome in ALL Survivors
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Sheba Medical Center (Other Government)
Responsible Party: Dr. Yael Weintraub, Sheba Medical Cener
Other Study IDs: SHEBA-07-4861-YW-CTIL
Record Dates: First submitted 2007-11-30; First posted 2007-12-03 (Estimated); Last update posted 2007-12-03 (Estimated); Status verified 2007-11

CONDITIONS: Leukemia; Metabolic Syndrome X
Keywords: adipocytokines; inflammatory markers; cardiovascular disease; diabetes mellitus; Leptin
MeSH Terms: conditions — Leukemia; Metabolic Syndrome; Cardiovascular Diseases; Diabetes Mellitus | interventions — DNA

STUDY DESIGN:
Observational Model: Cohort
Biospecimen Retention: Samples Without DNA — Serum leptin, resistin ,adiponectin ,CRP, PAI ,TNF-α, IL-6 will be taken as part of initial blood test screening in patients following an overnight fast. Adiponectin and leptin levels will be determined by RIA (Linco, St. Charles, MO), Insulin, will be determined by chemiluminescent immunometric method (Immulite 2000, Diagnostic Products Corporation, Los Angeles, CA).
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 1: ALL survivors 5 years after completion of treatment, during routine medical follow up
  Interventions: Other: sample without DNA

INTERVENTIONS:
Other: sample without DNA — family history, anthropometric measurements and blood sampling

SUMMARY:
Background: Acute Lymphoblastic Leukemia (ALL) is the most common malignancy in children. It accounts for 25% of all childhood cancers. Peak incidence occurs between 2 to 5 years of age. Modern treatment regimens have improved cure rates from virtually zero (in the 1950's) to current overall survival rates of approximately 80%.The high survival rates have introduced us to novel medical problems as a consequences of the different treatment regimens. No single treatment modality exists today but rather several treatment protocols are accepted worldwide. As such, the population of the childhood ALL survivors differ in their toxic exposure: cranial & spinal radiotherapy, intrathecal and/or systemic chemotherapy and bone marrow transplantation .As the survival rates grow, there are more young adult ALL survivors worldwide susceptible to these late effects of treatment.

Numerous reports have pointed out that this particular group is at increased risk to develop cardiovascular disease (CVD) and diabetes (MS). The metabolic syndrome, i.e hypertension, dyslipidemia, impaired glucose metabolism and obesity, occurs at a younger age than the general population.

Adipocytokines, mediators secreted by adipose tissue, play an important role in the regulation of carbohydrates and lipid metabolism.Changes in serum adipokine levels precede the clinical symptoms.

We aim to identify and assess prevalence of the MS in ALL survivors. We aim to characterize the population at risk to develop DM and CVD prior to overt clinical disease. Characterization will be done by measuring serum adipocytokines and inflammatory cytokine profiles .Biochemical characterization of the group at risk will enable us to intervene in the preventive stage in the future.

ELIGIBILITY:
Inclusion Criteria:

* ALL diagnosis
* five years after completion of treatment
* leukemia free during research

Exclusion Criteria:

* ongoing chemotherapy and radiotherapy

Ages: 6 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Hematoncological pediatric clinic
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2008-01; Study Completion 2008-12 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Yael Weintraub, MD, Principal Investigator — Tel Aviv University

REFERENCES:
- [Background] Eckel RH, Grundy SM, Zimmet PZ. The metabolic syndrome. Lancet. 2005 Apr 16-22;365(9468):1415-28. doi: 10.1016/S0140-6736(05)66378-7. PMID 15836891
- [Background] Alberti KG, Zimmet P, Shaw J; IDF Epidemiology Task Force Consensus Group. The metabolic syndrome--a new worldwide definition. Lancet. 2005 Sep 24-30;366(9491):1059-62. doi: 10.1016/S0140-6736(05)67402-8. No abstract available. PMID 16182882
- [Background] Cook S, Weitzman M, Auinger P, Nguyen M, Dietz WH. Prevalence of a metabolic syndrome phenotype in adolescents: findings from the third National Health and Nutrition Examination Survey, 1988-1994. Arch Pediatr Adolesc Med. 2003 Aug;157(8):821-7. doi: 10.1001/archpedi.157.8.821. PMID 12912790
- [Background] Taskinen M, Saarinen-Pihkala UM, Hovi L, Lipsanen-Nyman M. Impaired glucose tolerance and dyslipidaemia as late effects after bone-marrow transplantation in childhood. Lancet. 2000 Sep 16;356(9234):993-7. doi: 10.1016/S0140-6736(00)02717-3. PMID 11041401
- [Background] Gurney JG, Ness KK, Sibley SD, O'Leary M, Dengel DR, Lee JM, Youngren NM, Glasser SP, Baker KS. Metabolic syndrome and growth hormone deficiency in adult survivors of childhood acute lymphoblastic leukemia. Cancer. 2006 Sep 15;107(6):1303-12. doi: 10.1002/cncr.22120. PMID 16894525
- [Background] Mohn A, Di Marzio A, Capanna R, Fioritoni G, Chiarelli F. Persistence of impaired pancreatic beta-cell function in children treated for acute lymphoblastic leukaemia. Lancet. 2004 Jan 10;363(9403):127-8. doi: 10.1016/S0140-6736(03)15264-6. PMID 14726167
- [Background] Razzouk BI, Rose SR, Hongeng S, Wallace D, Smeltzer MP, Zacher M, Pui CH, Hudson MM. Obesity in survivors of childhood acute lymphoblastic leukemia and lymphoma. J Clin Oncol. 2007 Apr 1;25(10):1183-9. doi: 10.1200/JCO.2006.07.8709. PMID 17401007
- [Background] Kourti M, Tragiannidis A, Makedou A, Papageorgiou T, Rousso I, Athanassiadou F. Metabolic syndrome in children and adolescents with acute lymphoblastic leukemia after the completion of chemotherapy. J Pediatr Hematol Oncol. 2005 Sep;27(9):499-501. doi: 10.1097/01.mph.0000181428.63552.e9. PMID 16189445
- [Background] Oeffinger KC, Buchanan GR, Eshelman DA, Denke MA, Andrews TC, Germak JA, Tomlinson GE, Snell LE, Foster BM. Cardiovascular risk factors in young adult survivors of childhood acute lymphoblastic leukemia. J Pediatr Hematol Oncol. 2001 Oct;23(7):424-30. doi: 10.1097/00043426-200110000-00007. PMID 11878576
- [Background] Koerner A, Kratzsch J, Kiess W. Adipocytokines: leptin--the classical, resistin--the controversical, adiponectin--the promising, and more to come. Best Pract Res Clin Endocrinol Metab. 2005 Dec;19(4):525-46. doi: 10.1016/j.beem.2005.07.008. PMID 16311215
- [Background] Pui CH, Cheng C, Leung W, Rai SN, Rivera GK, Sandlund JT, Ribeiro RC, Relling MV, Kun LE, Evans WE, Hudson MM. Extended follow-up of long-term survivors of childhood acute lymphoblastic leukemia. N Engl J Med. 2003 Aug 14;349(7):640-9. doi: 10.1056/NEJMoa035091. PMID 12917300